CLINICAL TRIAL: NCT05799469
Title: A Single-arm Exploratory Clinical Study of Envafolimab With Chemoradiotherapy for Women With Locally Advanced Cervical Cancer
Brief Title: Study of Chemoradiotherapy With Envafolimab For The Treatment of Locally Advanced Cervical Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Principal Investigator, Qi Zhou, Professor, Chongqing University Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-CC-001
Record Dates: First submitted 2023-03-14; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Locally Advanced Cervical Cancer
Keywords: Cervical Cancer; Local advanced; Concurrent chemoradiotherapy; Immune checkpoint inhibitors
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — envafolimab; Cisplatin; Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): Participants receive envafolimab 150 mg subcutaneously (SC) on Day 1 of each week cycle (QW) for 8 cycles followed by envafolimab 300 mg SC on Day 1 of each 3-week cycle (Q3W) until disease progression, intolerable toxicity, investigator determines that the participant cannot continue to benefit, withdraws informed consent, or envafolimab treatment over 2 years. During the QW dosing period of envafolimab, participants receive concurrent chemoradiotherapy. The standard of care chemoradiotherapy regimen includes cisplatin 40 mg/m^2 IV once per week (QW) for 5 or 6 weeks plus external beam radiotherapy (EBRT) followed by brachytherapy with minimum total radiotherapy dose of 45 Gray Units (Gy)with the total duration of radiation treatment not to exceed 56 days.
  Interventions: Drug: Envafolimab; Drug: Cisplatin; Radiation: External Beam Radiotherapy (EBRT); Radiation: Brachytherapy (BT)

INTERVENTIONS:
Drug: Envafolimab — SC
  Other Names: KN035
Drug: Cisplatin — IV infusion
Radiation: External Beam Radiotherapy (EBRT) — 45-50.4Gy
Radiation: Brachytherapy (BT) — Performed according to clinically required dose

SUMMARY:
This is a single-arm, single-center, exploratory study, the purpose of this study is to evaluate the efficacy and safety of envafolimab combined with Chemoradiotherapy in participants with locally advanced cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* The subject voluntarily joins this study and is able to sign the informed consent form with good compliance;
* Female aged 18-75 years (at the time of signing the informed consent);
* ECOG score of 0-1 within 7 days prior to first study intervention dose;
* Expectation of life ≥ 12 weeks;
* Locally advanced squamous cell carcinoma , adenocarcinoma or adenosquamous -carcinoma of the cervix confirmed by pathological histological or clinical diagnosis according to cervical cancer F IGO stage (2018 version) as I B3 , IIA2 , IIB , I II-IVA stage ;
* Pathological specimens (≥ 18 eligible tissue sections) may be provided for biomarker testing;
* No prior surgery for cervical cancer (excluding staging surgery), radiotherapy, chemotherapy, systemic therapy (including investigational agents), or immunotherapy ;
* At least 1 measurable cervical lesion or metastatic lymph node meeting RECIST1.1 target lesion criteria by CT scan or MRI within 28 days prior to treatment;
* Adequate major organ function meeting the following criteria:

  1. Hematology (need not be transfused within 14 days and hematopoietic stimulating factor drugs within 7 days without correction testing): hemoglobin (Hb) ≥ 90 g/L; absolute neutrophil count (ANC) ≥ 1.5 × 109/L; platelets (PLT) ≥ 80 × 109/L;
  2. Biochemistry: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; serum total bilirubin (TBIL) ≤ 1.5 × ULN (in subjects with Gilbert 's syndrome, ≤ 3 × ULN); serum creatinine (Cr) ≤ 1.5 × ULN, or creatinine clearance ≥ 60 mL/min;
  3. Coagulation function: activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT) ≤ 1.5 × ULN;
  4. Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ 50%;
  5. Thyroid function is normal，defined as thyroid stimulating hormone (TSH) within normal limits. If baseline TSH is out of normal range, subjects with total T3 (or FT3) and FT4 within normal range can also be enrolled;
  6. Adequate organ function as judged clinically appropriate for the study by the physician.
* Subjects of childbearing potential must use adequate contraception during this study and for 120 days after the end of the study, have a negative serum pregnancy test within 7 days prior to study enrollment, and must be non-lactating.

Exclusion Criteria:

* Patients who had or currently had other malignant tumors within 3 years prior to the start of study treatment;
* Inability to perform (complete) brachytherapy due to anatomy, tumor shape, contraindications, etc.;
* Grade ≥ 1 unresolved toxicity due to any prior therapy (according to National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events Version 5.0 [CTCAE 5.0]);
* Subjects with any severe and/or uncontrolled disease. Including:

  1. Unsatisfactory blood pressure control (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg);
  2. Patients with ≥ Grade 2 myocardial ischemia or myocardial infarction, arrhythmia (QTc ≥ 470 ms) and ≥ Grade 2 congestive heart failure (New York Heart Association [NYHA] classification);
  3. Active or uncontrolled serious infection (≥ CTCAE Grade 2 infection);
  4. Cirrhosis, active hepatitis * ; * active hepatitis (hepatitis B reference: HBsAg positive, and HBV DNA test value more than the upper limit of normal; hepatitis C reference: HCV antibody positive, and HCV viral titer test value more than the upper limit of normal) ; patients with previous HBV infection or cured HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and the absence of HBsAg) are eligible; among patients with positive HCV antibody, patients can participate in this study only when HCV RNA is negative by polymerase chain reaction (PCR); Note: subjects with positive HBsAg or positive anti-HBc or hepatitis C，who are eligible for inclusion need continuous antiviral treatment to prevent virus activation ;
  5. Previous (non infectious) pneumonia/interstitial lung disease still requires steroid treatment or currently has (non infectious) lung disease;
  6. Active syphilis;
  7. Patients with renal failure requiring hemodialysis or peritoneal dialysis;
  8. Patients with a history of immunodeficiency, including HIV positive or suffering from other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
* Poorly controlled diabetes (fasting blood glucose [FBG] > 10 mmol/L);
* Urine routine showed urine protein ≥ + +, and confirmed 24-hour urine protein > 1.0g;
* Patients who received major surgical treatment or significant traumatic injury within 28 days prior to the start of study treatment; or had wounds or fractures that were not healed for a long time;
* Severe arterial/venous thrombotic events such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis and pulmonary embolism within 6 months before the start of study treatment;
* Patients who have a history of psychotropic substance abuse and cannot quit or have mental disorders;
* Study treatment related:

  1. History of live vaccination 28 days prior to start of study treatment or planned live vaccination during the study;
  2. Patients who have experienced severe hypersensitivity reactions after using monoclonal antibodies;
  3. Active autoimmune disease requiring systemic therapy (eg, use of therapeutic drugs, corticosteroids, or immunosuppressive agents) within 2 years prior to start of study treatment, with the exception of alternative therapies (eg, thyroxine, insulin, or physiologic corticosteroids for adrenal or pituitary insufficiency);
  4. Diagnosed with immunodeficiency or receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy (prednisone at a dose > 10 mg/day or other equivalent efficacy physiological dose hormone) and continued to use within 2 weeks before the first study dose;
  5. Patients with a history of active tuberculosis;
* Participating or participating in other clinical investigators;
* Patients who are unable to comply with the trial protocol or cooperate with follow-up according to the investigator 's judgment;
* Patients with a history of severe allergy;
* Known hypersensitivity to active ingredients or excipients of the study drug, such as envafolimab and cisplatin;
* Subjects who have concomitant diseases that, in the investigator 's judgment, would seriously jeopardize the subject' s safety or affect the completion of the study, or who are considered unsuitable for enrollment for other reasons.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) at Month 24 as Assessed by the Investigator | The cut-off date is event-driven and estimated to be approximately 48 months.
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. PFS data will be cumulated to a certain cut-off date and the analysis will be performed via Kaplan-Meier approach to estimate the PFS rate at Month 24 using the entire PFS data up to the cut-off date.

SECONDARY OUTCOMES:
Objective Response Rate(ORR) | Up to 2 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR per RECIST v1.1.
Duration of response (DoR) | Up to 2 years
  The DoR is defined as the time from first response to disease progression or death in the absence of disease progression. First response was defined as first CR or PR was achieved. DoR will be summarized for responding patients and DoR rates (%) at 12, 24, and 36 months will be provided.
Progression-Free Survival (PFS) at Month 12/36 | The cut-off date is event-driven and estimated to be approximately 48 months.
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. PFS data will be cumulated to a certain cut-off date and the analysis will be performed via Kaplan-Meier approach to estimate the PFS rate at Month 12/36 using the entire PFS data up to the cut-off date.
Overall Survival (OS) at Month 12/24/36 | The cut-off date is event-driven and estimated to be approximately 48 months.
  OS is the time from randomization to death due to any cause. OS data will be cumulated to a certain cut-off date and the analysis will be performed via Kaplan-Meier approach to estimate the OS rate at Month 12/24/36 using the entire OS data up to the cut-off date.
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Global Health Status Score and Physical Function Score. | Baseline and up to approximately 48 months
  The EORTC QLQ-C30 is a questionnaire that rates the overall quality of life in cancer participants. The first 28 questions use a 4-point scale (1=not at all to 4=very much) for evaluating function (physical, role, social, cognitive, emotional), symptoms (diarrhea, fatigue, dyspnea, appetite loss, insomnia, nausea/vomiting, constipation, and pain) and financial difficulties. The last 2 questions use a 7-point scale (1=very poor to 7=excellent) to evaluate overall health and quality of life. Global scores are converted to a score of 0 to 100, with a higher score indicating improved health status. The change from baseline in EORTC QLQ-C30 score will be presented.
Change from Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Symptom Specific Scale for Cervical Cancer (EORTC QLQ-CX24) Score. | Baseline and up to approximately 48 months
  The EORTC QLQ-CX24 is a questionnaire that rates the symptoms common to women with cervical cancer and evaluates the impact of disease and/or treatments. The 24 items use a 4-point scale (1=not at all to 4=very much) and are classified into 3 multi-item scales, 11 items with symptom experience, 3 items with body image, and 4 items with sexual/ vaginal functioning. The other items of the questionnaire are lymphedema, peripheral neuropathy, menopausal symptom, sexual worry, sexual activity, and sexual enjoyment. The change from baseline in EORTC QLQ-CX24 score will be presented.
Number of participants with adverse events (AEs) | Up to approximately 48 months
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Qi Zhou, PhD, Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- Chongqing university Cancer Hospital, Chongqing, CHN, China

IPD SHARING:
Plan to Share IPD: No